CLINICAL TRIAL: NCT02232958
Title: The Effect of Hyperbaric Oxygen on the Functional Connectivity of Resting State Neural Networks in Patients With Cerebral Small Vessel Disease
Brief Title: Effect of HBO on Functional Connectivity of Resting State Networks in Patients With Cerebral Small Vessel Disease
Acronym: HBO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funds depleted and Ilness of Principal Investigator
Sponsor: St. Luke's Hospital, Chesterfield, Missouri (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, John Davidson, Professor of Clinical Medicine Washington University School of Medicine, St. Luke's Hospital, Chesterfield, Missouri
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #2014.011
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Encephalopathy; White Matter Hyperintensities; Impaired Oxygen Delivery
Keywords: Hyperbaric Oxygen; Small Vessel Disease of the Brain; Impaired Brain Circuit Connections
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperbaric Oxygen treatment (Experimental): administration of 100% Oxygen at 2 Atmospheres Absolute for 1 hour 1 daily, 5 days a week for 2 weeks
  Interventions: Other: Hyperbaric Oxygen Treatment

INTERVENTIONS:
Other: Hyperbaric Oxygen Treatment — Patients are placed in a special chamber in which the pressure is gradually increased up to the desired pressure with 100% Oxygen and the patient is kept at that pressure for one hour. Then the Oxygen flow is slowly reduced until the patient has been returned to one atmosphere of pressure.

SUMMARY:
The purpose of this study is to extend our previous work, in which we demonstrated an increase in the internal and cross network connectivity of resting state neural networks in patients with cerebral small vessel disease by treatment with hyperbaric oxygen, to at least 20 more individuals.

DETAILED DESCRIPTION:
Patients without contraindications to Hyperbaric Oxygen treatment or magnetic resonance imaging who exhibit white matter hyper-intensities on MRI will be recruited to have a functional MRI followed by10 hyperbaric oxygen treatments at 2 ATA for one hour. These treatments will be done once daily, from Monday through Friday, on 2 consecutive weeks. 4-6 weeks later, they have a repeat fMRI. These fMRI's will be analyzed regarding any changes in the resting state connectivity of various circuits.

ELIGIBILITY:
Inclusion Criteria: Over 50 years of age White Matter Hyperintensities on MRI @ or more symptoms and/or neurological impairments e.g. gait disturbances,disequilibrium, decline in cognitive function, upper motor neuron deficit, dysmetria, hyper-refexia or unilateral increase in motor tone -

Exclusion Criteria: Contraindications to hyperbaric oxygen therapy e.g. pulmonary emphysema or bullae, claustrophobiia, seizure diorder Inability of the patient to tolerate pressurization e.g. Eustachian tube dysfunction Stroke within the previous 6 months Extreme cognitive impairment Major depression Other uncontrolled co-morbidities, e.g. diabetes, hypertension, thyroid disorders, carotid artery stenosis (>70%), renal or hepatic dysfunction History of brain tumor, head trauma, electric shock therapy, brain irradiation History of migraine headaches

-

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Evidence of an increase in the connectivity of resting state neural networks after treatment with hyperbaric oxygen | 4-6 weeks after treatment
  Patients with small vessel disease of the brain will be treated with 10 hyperbaric oxygen sessions for 1 hour at 2 atmospheres absolute over the course of 2 weeks. Functional connectivity MRIs will be obtained 4-6 weeks after these sessions for comparison with those obtained before hyperbaric oxygen exposure

SECONDARY OUTCOMES:
an improvement on the NIH Neurobehavioral scale compared to the one done before hyperbaric oxygen | 4-6 weeks
  NIH Neurobehavioral evaluations be obtained 4-6 weeks after exposure to 10 hyperbaric oxygen sessions of 1 hour at 2 atmospheres delivered over a period of 2 weeks. These will be compared to evaluations obtained prior to hyperbaric oxygen treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John D. Davidson, MD, Principal Investigator — St. Luke's Hospital St. Louis & Washington University Medical School
Locations (3):
- United States (3):
  - St. Luke's Hospital, Chesterfield, Missouri
  - St. Luke's Hospital, St Louis, Missouri
  - Mallinckrodt Institute of Radiology/Washington University Medical School, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No